CLINICAL TRIAL: NCT03655418
Title: "Jag Vill, Jag Kan, Jag törs!" Implementation and Effect Study of a Method to Promote Child Resilience
Brief Title: Implementation and Evaluation of RESCUR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: IOGT-NTO's Junior Association (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Rescur_Goteborg
Record Dates: First submitted 2018-08-21; First posted 2018-08-31 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Resilience

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The prevention program RECUR will be administered.
  Interventions: Other: Resilience Curriculum (RESCUR)
- Waitlist control (No Intervention): The prevention program RECUR will be administered after a year of waiting.

INTERVENTIONS:
Other: Resilience Curriculum (RESCUR) — The method of the present project, developed by experts in Europe, concerns giving children their own self-empowerment, strengthening protective factors, and, in the long run, their resilience. In Sweden, the material has been named "Jag vill, jag kan, jag törs!".
  The methodology that will be further developed and evaluated in this project is called RESCUR (the resilience curriculum) aimed at increasing children's resilience, i.e., children's ability to cope with crises, changes and stressors without falling apart. The method is rooted in research on human resilience.
  Arms: Intervention

SUMMARY:
This research program aims to investigate the implementation and effects of a theoretical promising prevention method developed in a European research collaboration within a Comenius project (2012-2015) between 6 European universities (in Malta, Italy, Greece, Croatia, Portugal and Sweden) with the purpose of enhancing European children's resilience.

RESCUR in Sweden is a RCT study of the Resilience Curriculum (RESCUR) that is taking place in Sweden 2017-2019. The Swedish name is "Jag vill, jag kan, jag törs!". The study is performed by Junis, IOGT-NTO's Junior Association, in conjunction with researchers at Göteborg, Umeå and Stockholm Universities and is being funded by the Public Health Agency of Sweden.

Around, 1,000 children of the ages 7-12 will, through their schools and associations, or via groups in social services, be made acquainted with the material The children will learn and practice Mindfulness activities, storytelling activities, group discussions and much more, all designed to strengthen protective factors and increase their resilience. The program also involves parents taking part in the work to reinforce children's protective factors.

Based on the work with groups of children, an effectiveness study including at children aged 7-12 in school classes, with randomized and controlled pre- and post-measurements, self-rating questionnaires and group observations takes place. The program will also be implemented in a non-governmental organization and in groups in social services. The study also investigates the forms of implementation

DETAILED DESCRIPTION:
This research program aims to investigate the implementation and effects of a theoretical promising prevention method developed in a European research collaboration within a Comenius project (2012-2015) between 6 European universities (in Malta, Italy, Greece, Croatia, Portugal and Sweden) with the purpose of enhancing European children's resilience.

RESCUR in Sweden is a RCT study of the Resilience Curriculum (RESCUR) that is taking place in Sweden 2017-2019. The Swedish name is "Jag vill, jag kan, jag törs!". The study is performed by Junis, IOGT-NTO's Junior Association, in conjunction with researchers at Göteborg, Umeå and Stockholm Universities and is being funded by the Public Health Agency of Sweden.

The primary aim is to strengthen protective factors and promote childhood life changes for 7-12 years who are relatives of people with addiction problems and to contribute to the support that Swedish society gives these children. This means a preventive intervention targeted towards those who have an increased risk of developing addiction problems and other problems that are consequences of their situation. A secondary aim at the universal level is to promote protective factors among children of the same ages, and to prevent the development of drug addiction in among children.

In order to increase our chances of achieving the aims, we are implementing the project as a collaboration between practitioners and researchers. Our aim is also to increase the relevance of the project as well as the development of knowledge and improve practical implementation. Moreover, this can also provide an increased opportunity to disseminate experience also to other groups and activities after the method has been tested and evaluated based on the Swedish context and in the three priority areas - social services, a NGO and schools.

The research includes five research questions:

1. How can participants in the implementation of the program be recruited?
2. How can leaders be supported to enable the implementation of the high-quality program?
3. What is the significance of the program for children's development and mental health?
4. Does the program work differently for different groups in relation to gender, social background, place of residence and age?
5. Does the intervention work differently at a universal, selective or indicative level?

Research questions will be studied through an implementation evaluation, using self-assessment forms, interviews and observations using an established "checklist", as well as through an impact assessment, which has a randomized, controlled pre-post design, and in which self-reports, interviews and adult reports of testing instruments are used. Our main target group for research is children who are seven to twelve years in Sweden and who are in one of the organizations school, social services or the value-based organization IOGT-NTO's Junior Association, Junis. A secondary target is the deliverers.

The project is divided into three phases. The first phase involved planning and a preliminary study including the application for research ethics committee (first year). We started the project, formed a project team and appointed a project manager, worked on the manuals to make them more user-friendly, informed and marketed the project to organizations and policy-makers, recruited participants for the evaluation, finalized the project and research plan, including all measuring instruments. The ethical review board approved the research project.

The project is based on close cooperation between Junis and the research group with a clear division of work and responsibility. The purpose of Junis's activities is to provide health promotion for children aged 7-15 years in an encouraging environment where the child's self-esteem and self-confidence grow together with secure and safe adults. The organization is be responsible for planning and implementing the program in all groups. The research group is responsible for the scientific study of implementation and effects of the program for the participants in groups and school classes that are part of intervention and control groups. The research is a randomized, controlled, longitudinal survey of the RESCUR program. This means a baseline measurements before the intervention begins and follow up at six months, one year and then two years.

The second phase involves implementing the program "Jag vill, jag lkan, jag törs!" (RESCUR) in Junis' group activities, in groups through social services and in school classes in different municipalities and spread across the country (ie. in different housing areas). The third phase involves analysis and reporting from the project's implementation and its effects.

The project will be carefully evaluated from two perspectives, implementation and impact. We will study the implementation through both self-assessment forms, reported by group leaders when the program has been used for half a year, and observations made according to a formalized checklist. The implementation of the method is fundamental in order to properly evaluate the effect of the method, which is the second part of the evaluation of the project. At the same time, we are also interested in directly studying the extent to which it is possible to implement the method as intended.

The effect of the method on protective factors and resilience will be measured via a randomized, controlled pre-post follow-up design with two types of groups. We will study the effect of the method from both a statistical significance perspective and a practical relevance perspective [62]. We will use our waiting list to create a control condition. The waiting list group is offered to start the intervention one year after base line measurements has taken place. We make a pre-measurement before the intervention begins among the participants, even adult reports will be collected, as well as measurements after one semester, one year and two years.

The controlled study has three different arms. In the case of schools, we have cluster randomize participants to one of two conditions, (A) intervention schools or (B) waiting list or control schools. Randomization has been done at school level. Thereafter, the baseline measurements were performed in both conditions, and after that, the intervention group began the action and measurements were made as described above (Table 1). One year after the baseline measurement intervention group (A) the waiting list group began the program. Measurements are finally made a year later.

In the case of Junis's groups, it was not feasible to do a cluster randomization at the managerial level as the involvement of local chapters was more difficult to achieve. The groups will be led by regular June volunteers.

As for the social service group, we will have the same arrangement and no waiting-list control condition. Here, a new round of groups is planned in the second year. On the other hand, we will have a follow-up measurement of the first wave's intervention groups in year 3 for both Junis and the social services groups. The groups will be run by social workers.

A calculation of the statistical power has been made for the interventions. In the universal intervention, an effect size of d = 0.3 and a power of 0.8 and the corresponding statistics are expected to test a group size of 176 in each group. The recruitment of schools for the evaluation of RESCUR has been completed. The data collection sites are recruited from different part of Sweden as well as in both urban and rural areas.

ELIGIBILITY:
* Child is between the ages of 7 and 12 years.
* Child is part of a school class, a social service group, or an NGO group that has implemented the RESCUR program.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 750 (Actual)
Dates: Start 2017-01-04 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Child and Youth Resilience Measure (CYRM-28) | 0-12 months
  A primary outcome measure in the effectiveness study is the "Child and Youth Resilience Measure" developed by Ungar et al (Liebenberg, Ungar & Van De Vijver, 2012) in Canada. The CYRM-28 measures aspects of resilience (i.e., developmental strenghts and assests) in children's characteristics and in their environment using 28 items that are reported on 5-point Likert scales by teachers or parents. Higher scores represent higher resilience. Total scores and mean values of the included items will be calculated. Higher scores at posttest compared to pretest and in the intervention group compared to the control group, indicate that the intervention was succesful.

SECONDARY OUTCOMES:
Strengths and difficulties questionnaire (SDQ) | 0-12 months
  The Strength and Difficulties questionnaire (SDQ, Goodman, 1997) measures children's psychological attributes including prosocial behavior (5 items), emotional symptoms (5 items), conduct problems (5 items), hyperactivity/inattention (5 items), and peer relationship problems using 25 items that teachers or parents answer on 3-point Likert scales. Total scores and mean values of the included items for each subscale will be calculated. The higher the score on one subscale, the more children have of that type of behavior. Higher prosocial behavior, and lower scores on the other subscales at posttest compared to pretest, and in the onterventiongroup compared to the control group, indicate that the intervention was successful.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lilja JL, Kimber B, Eriksson C, Henriksson B, Skoog T. Does the Delivery System Matter? The Scaling-Out of a School-Based Resilience Curriculum to the Social Services Sector. Front Psychiatry. 2021 May 4;12:578048. doi: 10.3389/fpsyt.2021.578048. eCollection 2021. PMID 34017270
- [Derived] Eriksson C, Kimber B, Skoog T. Design and implementation of RESCUR in Sweden for promoting resilience in children: a study protocol. BMC Public Health. 2018 Nov 12;18(1):1250. doi: 10.1186/s12889-018-6145-7. PMID 30419888